CLINICAL TRIAL: NCT04088630
Title: Fingolimod as a Treatment of Cerebral Edema After Intracerebral Hemorrhage
Acronym: FITCH
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00060619; UL1TR001420 (NIH)
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-02

CONDITIONS: Intracerebral Hemorrhage; Cerebral Edema; Stroke Hemorrhagic; Intracerebral Hemorrhage, Hypertensive; Intracerebral Hemorrhage Intraparenchymal
Keywords: Fingolimod; Neurologic Deficits; Brain Injury; Stroke; Intracerebral hemorrhage; Neuroimmunomodulation
MeSH Terms: conditions — Cerebral Hemorrhage; Brain Edema; Hemorrhagic Stroke; Intracranial Hemorrhage, Hypertensive; Neurologic Manifestations; Brain Injuries; Stroke | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled pilot trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Consented participants who can be administered an oral drug will be allocated to Fingolimod or Placebo study groups using a computer-based random number-generating allocation. Consented participants who are unable to be administered the oral drug or placebo are assigned to the open-label group. The study pharmacist will be the only member of the study to be unblinded to oral fingolimod or placebo randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fingolimod (Experimental): In addition to Standard of care treatment, those participants randomized to the fingolimod group will receive a single dose of 0.5 mg oral fingolimod within 24 hours of symptom onset.
  Interventions: Drug: Fingolimod
- Placebo Control (Placebo Comparator): In addition to Standard of care treatment, those participants randomized to the control group will receive a single dose placebo pill within 24 hours of symptom onset
  Interventions: Drug: Placebo
- Open-label Fingolimod (Experimental): In addition to standard of care treatment,10 subjects who are unable to be administered oral medication will be assigned to the open-label group who will receive a single dose of 0.5 mg oral fingolimod within 24 hours of symptom onset to assess feasibility of administration through NGT or Dobhoff tube.
  Interventions: Drug: Open-label Fingolimod

INTERVENTIONS:
Drug: Fingolimod — A single dose of 0.5 mg oral fingolimod within 24 hours of symptom onset
  Arms: Fingolimod
Drug: Placebo — A single oral placebo pill within 24 hours of symptom onset
  Arms: Placebo Control
Drug: Open-label Fingolimod — A single dose of 0.5 mg fingolimod through an NGT or Dobhoff tube within 24 hours of symptom onset
  Arms: Open-label Fingolimod

SUMMARY:
The purpose of this study is to test the safety and effectiveness of a single dose of fingolimod in patients with primary spontaneous intracerebral hemorrhage (ICH).

DETAILED DESCRIPTION:
This is a double-blinded, placebo-controlled pilot trial of fingolimod in patients with primary spontaneous intracerebral hemorrhage. Eligible participants will be allocated to study groups using fixed allocation randomization and a computer-based random number-generating allocation. For those patients who meet all inclusion criteria without exclusion criteria subjects will receive oral or nasogastric tube (NGT) or Dobhoff feeding tube administration of fingolimod versus placebo. Participants will be monitored at time of enrollment and days 1, 3 5, 7, and 14 (discharge dependent) by 2 blinded assessors (neuroscience subspecialists) and will receive standard of care for the duration of the study. After discharge from the hospital, participants will enter a follow up phase of 12 months, with clinic visits at 30±14 days, 90±14 days, 180±14 days, and 365±14 days. They will receive a standard of care neuroimaging at these follow up time-points and will be assessed with the pre-selected outcome assessments established by the NINDS Common Data Elements for Stroke.

ELIGIBILITY:
Inclusion Criteria:

Has given written informed consent to participate in the study in accordance with required regulations; if a participant is not capable of providing informed consent, written consent must be obtained from the participant's legally authorized representative (LAR). When the LAR is not available for consent, Docusign for econsent may be obtained.

Stated willingness to comply with all study procedures and availability for the duration of the study.

Men and non-pregnant women ages 18-80 years old Has a confirmed diagnosis of spontaneous supratentorial ICH. The presence of cerebellar ICH is exclusionary. Presence of hydrocephalus due to mass effect and cerebral edema is not exclusionary. If the patient has hydrocephalus requiring CSF drainage, an external ventricular drain will be placed as standard of care and will not be exclusionary.

Symptoms less than 24 hours prior to enrollment if all eligibility criteria are met. An unknown time of onset is exclusionary. Use the time the patient was last known to be well for patients that awaken from sleep with symptoms.

Has a GCS score ≥ 5 on presentation. Has a National Institutes of Health Stroke Scale (NIHSS) score ≥ 4 on presentation.

Maintenance of SBP < 200 mmHg at the time of enrollment and randomization. Historical Modified Rankin Scale score of 0-2.

Exclusion Criteria:

Men or women < 18 years old Incarcerated patients ICH known as a result of trauma. Primary intraventricular hemorrhage without significant intraparenchymal component.

Ruptured aneurysm, arteriovenous malformation (AVM), vascular anomaly, Moyamoya disease, hemorrhagic conversion of an ischemic infarct, recurrence of recent (< 1 year) hemorrhage, neoplasms diagnosed with radiographic imaging.

Patients with unstable mass or evolving intracranial compartment syndrome. Brainstem hemorrhage or irreversible impaired brain stem function (bilateral fixed, dilated pupils and extensor motor posturing), GCS ≤ 4.

Platelet count < 100,000; INR > 1.4. Any irreversible coagulopathy or known clotting disorder. Known history of Mobitz Type II second-degree or third-degree atrioventricular (AV) block or sick sinus syndrome.

Admission within the past 6 months for the following: myocardial infarction, unstable angina, stroke, decompensated heart failure requiring hospitalization, or Class III/IV heart failure.

Baseline QTc interval ≥500 ms. Current treatment with Class Ia or Class III anti-arrhythmic drugs. Implanted cardiac devices that are not compatible with the desired MRI sequences needed for the study (non-contrast T1, T2, SWI/GRE, and FLAIR sequences).

Abnormal liver function or liver failure. Active acute infection that is deemed by the Principal Investigator to be clinically significant.

Chronic viral or fungal infection. Active use of antineoplastic, immunosuppressive, or immunomodulating therapies. Leukopenia with a WBC < 2.0 x 109/L. Not expected to survive to the 365 day visit due to co-morbidities or is DNR/DNI status prior to randomization.

Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.

Concomitant enrollment in another interventional study. Inability or unwillingness of participant or legal guardian/representative to give written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Q Wolfe, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Qureshi AI, Mendelow AD, Hanley DF. Intracerebral haemorrhage. Lancet. 2009 May 9;373(9675):1632-44. doi: 10.1016/S0140-6736(09)60371-8. PMID 19427958
- [Background] van Asch CJ, Luitse MJ, Rinkel GJ, van der Tweel I, Algra A, Klijn CJ. Incidence, case fatality, and functional outcome of intracerebral haemorrhage over time, according to age, sex, and ethnic origin: a systematic review and meta-analysis. Lancet Neurol. 2010 Feb;9(2):167-76. doi: 10.1016/S1474-4422(09)70340-0. Epub 2010 Jan 5. PMID 20056489
- [Background] Fogelholm R, Murros K, Rissanen A, Avikainen S. Long term survival after primary intracerebral haemorrhage: a retrospective population based study. J Neurol Neurosurg Psychiatry. 2005 Nov;76(11):1534-8. doi: 10.1136/jnnp.2004.055145. PMID 16227546
- [Background] WRITING GROUP MEMBERS; Lloyd-Jones D, Adams RJ, Brown TM, Carnethon M, Dai S, De Simone G, Ferguson TB, Ford E, Furie K, Gillespie C, Go A, Greenlund K, Haase N, Hailpern S, Ho PM, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott MM, Meigs J, Mozaffarian D, Mussolino M, Nichol G, Roger VL, Rosamond W, Sacco R, Sorlie P, Roger VL, Thom T, Wasserthiel-Smoller S, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2010 update: a report from the American Heart Association. Circulation. 2010 Feb 23;121(7):e46-e215. doi: 10.1161/CIRCULATIONAHA.109.192667. Epub 2009 Dec 17. No abstract available. PMID 20019324
- [Background] Qureshi AI, Suri MF, Nasar A, Kirmani JF, Ezzeddine MA, Divani AA, Giles WH. Changes in cost and outcome among US patients with stroke hospitalized in 1990 to 1991 and those hospitalized in 2000 to 2001. Stroke. 2007 Jul;38(7):2180-4. doi: 10.1161/STROKEAHA.106.467506. Epub 2007 May 24. PMID 17525400
- [Background] Adeoye O, Broderick JP. Advances in the management of intracerebral hemorrhage. Nat Rev Neurol. 2010 Nov;6(11):593-601. doi: 10.1038/nrneurol.2010.146. Epub 2010 Sep 28. PMID 20877400
- [Background] Xi G, Keep RF, Hoff JT. Mechanisms of brain injury after intracerebral haemorrhage. Lancet Neurol. 2006 Jan;5(1):53-63. doi: 10.1016/S1474-4422(05)70283-0. PMID 16361023
- [Background] Ariesen MJ, Claus SP, Rinkel GJ, Algra A. Risk factors for intracerebral hemorrhage in the general population: a systematic review. Stroke. 2003 Aug;34(8):2060-5. doi: 10.1161/01.STR.0000080678.09344.8D. Epub 2003 Jul 3. PMID 12843354
- [Background] Broderick JP, Brott TG, Duldner JE, Tomsick T, Huster G. Volume of intracerebral hemorrhage. A powerful and easy-to-use predictor of 30-day mortality. Stroke. 1993 Jul;24(7):987-93. doi: 10.1161/01.str.24.7.987. PMID 8322400
- [Background] Mould WA, Carhuapoma JR, Muschelli J, Lane K, Morgan TC, McBee NA, Bistran-Hall AJ, Ullman NL, Vespa P, Martin NA, Awad I, Zuccarello M, Hanley DF; MISTIE Investigators. Minimally invasive surgery plus recombinant tissue-type plasminogen activator for intracerebral hemorrhage evacuation decreases perihematomal edema. Stroke. 2013 Mar;44(3):627-34. doi: 10.1161/STROKEAHA.111.000411. Epub 2013 Feb 7. PMID 23391763
- [Background] Mendelow AD, Gregson BA, Rowan EN, Murray GD, Gholkar A, Mitchell PM; STICH II Investigators. Early surgery versus initial conservative treatment in patients with spontaneous supratentorial lobar intracerebral haematomas (STICH II): a randomised trial. Lancet. 2013 Aug 3;382(9890):397-408. doi: 10.1016/S0140-6736(13)60986-1. Epub 2013 May 29. PMID 23726393
- [Background] Morgenstern LB, Hemphill JC 3rd, Anderson C, Becker K, Broderick JP, Connolly ES Jr, Greenberg SM, Huang JN, MacDonald RL, Messe SR, Mitchell PH, Selim M, Tamargo RJ; American Heart Association Stroke Council and Council on Cardiovascular Nursing. Guidelines for the management of spontaneous intracerebral hemorrhage: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2010 Sep;41(9):2108-29. doi: 10.1161/STR.0b013e3181ec611b. Epub 2010 Jul 22. PMID 20651276
- [Background] Babu R, Bagley JH, Di C, Friedman AH, Adamson C. Thrombin and hemin as central factors in the mechanisms of intracerebral hemorrhage-induced secondary brain injury and as potential targets for intervention. Neurosurg Focus. 2012 Apr;32(4):E8. doi: 10.3171/2012.1.FOCUS11366. PMID 22463118
- [Background] Zhou Y, Wang Y, Wang J, Anne Stetler R, Yang QW. Inflammation in intracerebral hemorrhage: from mechanisms to clinical translation. Prog Neurobiol. 2014 Apr;115:25-44. doi: 10.1016/j.pneurobio.2013.11.003. Epub 2013 Nov 26. PMID 24291544
- [Background] Wang J. Preclinical and clinical research on inflammation after intracerebral hemorrhage. Prog Neurobiol. 2010 Dec;92(4):463-77. doi: 10.1016/j.pneurobio.2010.08.001. Epub 2010 Aug 14. PMID 20713126
- [Background] Wang J, Dore S. Inflammation after intracerebral hemorrhage. J Cereb Blood Flow Metab. 2007 May;27(5):894-908. doi: 10.1038/sj.jcbfm.9600403. Epub 2006 Oct 11. PMID 17033693
- [Background] Aronowski J, Zhao X. Molecular pathophysiology of cerebral hemorrhage: secondary brain injury. Stroke. 2011 Jun;42(6):1781-6. doi: 10.1161/STROKEAHA.110.596718. Epub 2011 Apr 28. PMID 21527759
- [Background] Keep RF, Hua Y, Xi G. Intracerebral haemorrhage: mechanisms of injury and therapeutic targets. Lancet Neurol. 2012 Aug;11(8):720-31. doi: 10.1016/S1474-4422(12)70104-7. Epub 2012 Jun 13. PMID 22698888
- [Background] Boche D, Perry VH, Nicoll JA. Review: activation patterns of microglia and their identification in the human brain. Neuropathol Appl Neurobiol. 2013 Feb;39(1):3-18. doi: 10.1111/nan.12011. PMID 23252647
- [Background] Lawson LJ, Perry VH, Dri P, Gordon S. Heterogeneity in the distribution and morphology of microglia in the normal adult mouse brain. Neuroscience. 1990;39(1):151-70. doi: 10.1016/0306-4522(90)90229-w. PMID 2089275
- [Background] Xiong XY, Liu L, Yang QW. Functions and mechanisms of microglia/macrophages in neuroinflammation and neurogenesis after stroke. Prog Neurobiol. 2016 Jul;142:23-44. doi: 10.1016/j.pneurobio.2016.05.001. Epub 2016 May 7. PMID 27166859
- [Background] Wasserman JK, Zhu X, Schlichter LC. Evolution of the inflammatory response in the brain following intracerebral hemorrhage and effects of delayed minocycline treatment. Brain Res. 2007 Nov 14;1180:140-54. doi: 10.1016/j.brainres.2007.08.058. Epub 2007 Sep 5. PMID 17919462
- [Background] Taylor RA, Sansing LH. Microglial responses after ischemic stroke and intracerebral hemorrhage. Clin Dev Immunol. 2013;2013:746068. doi: 10.1155/2013/746068. Epub 2013 Oct 10. PMID 24223607
- [Background] Mracsko E, Veltkamp R. Neuroinflammation after intracerebral hemorrhage. Front Cell Neurosci. 2014 Nov 20;8:388. doi: 10.3389/fncel.2014.00388. eCollection 2014. PMID 25477782
- [Background] Kanazawa M, Ninomiya I, Hatakeyama M, Takahashi T, Shimohata T. Microglia and Monocytes/Macrophages Polarization Reveal Novel Therapeutic Mechanism against Stroke. Int J Mol Sci. 2017 Oct 13;18(10):2135. doi: 10.3390/ijms18102135. PMID 29027964
- [Background] Zhao H, Garton T, Keep RF, Hua Y, Xi G. Microglia/Macrophage Polarization After Experimental Intracerebral Hemorrhage. Transl Stroke Res. 2015 Dec;6(6):407-9. doi: 10.1007/s12975-015-0428-4. Epub 2015 Oct 7. No abstract available. PMID 26446073
- [Background] Lan X, Han X, Li Q, Yang QW, Wang J. Modulators of microglial activation and polarization after intracerebral haemorrhage. Nat Rev Neurol. 2017 Jul;13(7):420-433. doi: 10.1038/nrneurol.2017.69. Epub 2017 May 19. PMID 28524175
- [Background] Zhang Z, Zhang Z, Lu H, Yang Q, Wu H, Wang J. Microglial Polarization and Inflammatory Mediators After Intracerebral Hemorrhage. Mol Neurobiol. 2017 Apr;54(3):1874-1886. doi: 10.1007/s12035-016-9785-6. Epub 2016 Feb 19. PMID 26894396
- [Background] Hu X, Leak RK, Shi Y, Suenaga J, Gao Y, Zheng P, Chen J. Microglial and macrophage polarization-new prospects for brain repair. Nat Rev Neurol. 2015 Jan;11(1):56-64. doi: 10.1038/nrneurol.2014.207. Epub 2014 Nov 11. PMID 25385337
- [Background] Eggen BJ, Raj D, Hanisch UK, Boddeke HW. Microglial phenotype and adaptation. J Neuroimmune Pharmacol. 2013 Sep;8(4):807-23. doi: 10.1007/s11481-013-9490-4. Epub 2013 Jul 25. PMID 23881706
- [Background] Shichita T, Sakaguchi R, Suzuki M, Yoshimura A. Post-ischemic inflammation in the brain. Front Immunol. 2012 May 31;3:132. doi: 10.3389/fimmu.2012.00132. eCollection 2012. PMID 22833743
- [Background] Hendrix S, Nitsch R. The role of T helper cells in neuroprotection and regeneration. J Neuroimmunol. 2007 Mar;184(1-2):100-12. doi: 10.1016/j.jneuroim.2006.11.019. Epub 2007 Jan 2. PMID 17198734
- [Background] Kivisakk P, Mahad DJ, Callahan MK, Trebst C, Tucky B, Wei T, Wu L, Baekkevold ES, Lassmann H, Staugaitis SM, Campbell JJ, Ransohoff RM. Human cerebrospinal fluid central memory CD4+ T cells: evidence for trafficking through choroid plexus and meninges via P-selectin. Proc Natl Acad Sci U S A. 2003 Jul 8;100(14):8389-94. doi: 10.1073/pnas.1433000100. Epub 2003 Jun 26. PMID 12829791
- [Background] Arumugam TV, Granger DN, Mattson MP. Stroke and T-cells. Neuromolecular Med. 2005;7(3):229-42. doi: 10.1385/NMM:7:3:229. PMID 16247183
- [Background] Yilmaz G, Arumugam TV, Stokes KY, Granger DN. Role of T lymphocytes and interferon-gamma in ischemic stroke. Circulation. 2006 May 2;113(17):2105-12. doi: 10.1161/CIRCULATIONAHA.105.593046. Epub 2006 Apr 24. PMID 16636173
- [Background] Hurn PD, Subramanian S, Parker SM, Afentoulis ME, Kaler LJ, Vandenbark AA, Offner H. T- and B-cell-deficient mice with experimental stroke have reduced lesion size and inflammation. J Cereb Blood Flow Metab. 2007 Nov;27(11):1798-805. doi: 10.1038/sj.jcbfm.9600482. Epub 2007 Mar 28. PMID 17392692
- [Background] Liesz A, Suri-Payer E, Veltkamp C, Doerr H, Sommer C, Rivest S, Giese T, Veltkamp R. Regulatory T cells are key cerebroprotective immunomodulators in acute experimental stroke. Nat Med. 2009 Feb;15(2):192-9. doi: 10.1038/nm.1927. Epub 2009 Jan 25. PMID 19169263
- [Background] Zhou K, Zhong Q, Wang YC, Xiong XY, Meng ZY, Zhao T, Zhu WY, Liao MF, Wu LR, Yang YR, Liu J, Duan CM, Li J, Gong QW, Liu L, Yang MH, Xiong A, Wang J, Yang QW. Regulatory T cells ameliorate intracerebral hemorrhage-induced inflammatory injury by modulating microglia/macrophage polarization through the IL-10/GSK3beta/PTEN axis. J Cereb Blood Flow Metab. 2017 Mar;37(3):967-979. doi: 10.1177/0271678X16648712. Epub 2016 Jul 20. PMID 27174997
- [Background] Loftspring MC, McDole J, Lu A, Clark JF, Johnson AJ. Intracerebral hemorrhage leads to infiltration of several leukocyte populations with concomitant pathophysiological changes. J Cereb Blood Flow Metab. 2009 Jan;29(1):137-43. doi: 10.1038/jcbfm.2008.114. Epub 2008 Oct 1. PMID 18827833
- [Background] Guo FQ, Li XJ, Chen LY, Yang H, Dai HY, Wei YS, Huang YL, Yang YS, Sun HB, Xu YC, Yang ZL. [Study of relationship between inflammatory response and apoptosis in perihematoma region in patients with intracerebral hemorrhage]. Zhongguo Wei Zhong Bing Ji Jiu Yi Xue. 2006 May;18(5):290-3. Chinese. PMID 16700995
- [Background] Gelderblom M, Leypoldt F, Steinbach K, Behrens D, Choe CU, Siler DA, Arumugam TV, Orthey E, Gerloff C, Tolosa E, Magnus T. Temporal and spatial dynamics of cerebral immune cell accumulation in stroke. Stroke. 2009 May;40(5):1849-57. doi: 10.1161/STROKEAHA.108.534503. Epub 2009 Mar 5. PMID 19265055
- [Background] Gu L, Xiong X, Zhang H, Xu B, Steinberg GK, Zhao H. Distinctive effects of T cell subsets in neuronal injury induced by cocultured splenocytes in vitro and by in vivo stroke in mice. Stroke. 2012 Jul;43(7):1941-6. doi: 10.1161/STROKEAHA.112.656611. Epub 2012 Jun 7. PMID 22678086
- [Background] Theodorou GL, Marousi S, Ellul J, Mougiou A, Theodori E, Mouzaki A, Karakantza M. T helper 1 (Th1)/Th2 cytokine expression shift of peripheral blood CD4+ and CD8+ T cells in patients at the post-acute phase of stroke. Clin Exp Immunol. 2008 Jun;152(3):456-63. doi: 10.1111/j.1365-2249.2008.03650.x. Epub 2008 Apr 16. PMID 18422734
- [Background] Gao L, Lu Q, Huang LJ, Ruan LH, Yang JJ, Huang WL, ZhuGe WS, Zhang YL, Fu B, Jin KL, ZhuGe QC. Transplanted neural stem cells modulate regulatory T, gammadelta T cells and corresponding cytokines after intracerebral hemorrhage in rats. Int J Mol Sci. 2014 Mar 13;15(3):4431-41. doi: 10.3390/ijms15034431. PMID 24633197
- [Background] Mao LL, Yuan H, Wang WW, Wang YJ, Yang MF, Sun BL, Zhang ZY, Yang XY. Adoptive Regulatory T-cell Therapy Attenuates Perihematomal Inflammation in a Mouse Model of Experimental Intracerebral Hemorrhage. Cell Mol Neurobiol. 2017 Jul;37(5):919-929. doi: 10.1007/s10571-016-0429-1. Epub 2016 Sep 27. PMID 27678140
- [Background] Kappos L, Radue EW, O'Connor P, Polman C, Hohlfeld R, Calabresi P, Selmaj K, Agoropoulou C, Leyk M, Zhang-Auberson L, Burtin P; FREEDOMS Study Group. A placebo-controlled trial of oral fingolimod in relapsing multiple sclerosis. N Engl J Med. 2010 Feb 4;362(5):387-401. doi: 10.1056/NEJMoa0909494. Epub 2010 Jan 20. PMID 20089952
- [Background] Calabresi PA, Radue EW, Goodin D, Jeffery D, Rammohan KW, Reder AT, Vollmer T, Agius MA, Kappos L, Stites T, Li B, Cappiello L, von Rosenstiel P, Lublin FD. Safety and efficacy of fingolimod in patients with relapsing-remitting multiple sclerosis (FREEDOMS II): a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Neurol. 2014 Jun;13(6):545-56. doi: 10.1016/S1474-4422(14)70049-3. Epub 2014 Mar 28. PMID 24685276
- [Background] Groves A, Kihara Y, Chun J. Fingolimod: direct CNS effects of sphingosine 1-phosphate (S1P) receptor modulation and implications in multiple sclerosis therapy. J Neurol Sci. 2013 May 15;328(1-2):9-18. doi: 10.1016/j.jns.2013.02.011. Epub 2013 Mar 19. PMID 23518370
- [Background] Cohen JA, Chun J. Mechanisms of fingolimod's efficacy and adverse effects in multiple sclerosis. Ann Neurol. 2011 May;69(5):759-77. doi: 10.1002/ana.22426. PMID 21520239
- [Background] Chun J, Hartung HP. Mechanism of action of oral fingolimod (FTY720) in multiple sclerosis. Clin Neuropharmacol. 2010 Mar-Apr;33(2):91-101. doi: 10.1097/WNF.0b013e3181cbf825. PMID 20061941
- [Background] Chiba K. FTY720, a new class of immunomodulator, inhibits lymphocyte egress from secondary lymphoid tissues and thymus by agonistic activity at sphingosine 1-phosphate receptors. Pharmacol Ther. 2005 Dec;108(3):308-19. doi: 10.1016/j.pharmthera.2005.05.002. Epub 2005 Jun 13. PMID 15951022
- [Background] Lee CW, Choi JW, Chun J. Neurological S1P signaling as an emerging mechanism of action of oral FTY720 (fingolimod) in multiple sclerosis. Arch Pharm Res. 2010 Oct;33(10):1567-74. doi: 10.1007/s12272-010-1008-5. Epub 2010 Oct 30. PMID 21052934
- [Background] David OJ, Kovarik JM, Schmouder RL. Clinical pharmacokinetics of fingolimod. Clin Pharmacokinet. 2012 Jan 1;51(1):15-28. doi: 10.2165/11596550-000000000-00000. PMID 22149256
- [Background] Jin Y, Zollinger M, Borell H, Zimmerlin A, Patten CJ. CYP4F enzymes are responsible for the elimination of fingolimod (FTY720), a novel treatment of relapsing multiple sclerosis. Drug Metab Dispos. 2011 Feb;39(2):191-8. doi: 10.1124/dmd.110.035378. Epub 2010 Nov 2. PMID 21045201
- [Background] Zollinger M, Gschwind HP, Jin Y, Sayer C, Zecri F, Hartmann S. Absorption and disposition of the sphingosine 1-phosphate receptor modulator fingolimod (FTY720) in healthy volunteers: a case of xenobiotic biotransformation following endogenous metabolic pathways. Drug Metab Dispos. 2011 Feb;39(2):199-207. doi: 10.1124/dmd.110.035907. Epub 2010 Nov 2. PMID 21045200
- [Background] Kovarik JM, Schmouder R, Barilla D, Wang Y, Kraus G. Single-dose FTY720 pharmacokinetics, food effect, and pharmacological responses in healthy subjects. Br J Clin Pharmacol. 2004 May;57(5):586-91. doi: 10.1111/j.1365-2125.2003.02065.x. PMID 15089811
- [Background] Budde K, Schmouder RL, Brunkhorst R, Nashan B, Lucker PW, Mayer T, Choudhury S, Skerjanec A, Kraus G, Neumayer HH. First human trial of FTY720, a novel immunomodulator, in stable renal transplant patients. J Am Soc Nephrol. 2002 Apr;13(4):1073-1083. doi: 10.1681/ASN.V1341073. PMID 11912269
- [Background] Tham CS, Lin FF, Rao TS, Yu N, Webb M. Microglial activation state and lysophospholipid acid receptor expression. Int J Dev Neurosci. 2003 Dec;21(8):431-43. doi: 10.1016/j.ijdevneu.2003.09.003. PMID 14659994
- [Background] Okada T, Kajimoto T, Jahangeer S, Nakamura S. Sphingosine kinase/sphingosine 1-phosphate signalling in central nervous system. Cell Signal. 2009 Jan;21(1):7-13. doi: 10.1016/j.cellsig.2008.07.011. Epub 2008 Jul 22. PMID 18694820
- [Background] Melendez AJ. Sphingosine kinase signalling in immune cells: potential as novel therapeutic targets. Biochim Biophys Acta. 2008 Jan;1784(1):66-75. doi: 10.1016/j.bbapap.2007.07.013. Epub 2007 Aug 14. PMID 17913601
- [Background] Nayak D, Huo Y, Kwang WX, Pushparaj PN, Kumar SD, Ling EA, Dheen ST. Sphingosine kinase 1 regulates the expression of proinflammatory cytokines and nitric oxide in activated microglia. Neuroscience. 2010 Mar 10;166(1):132-44. doi: 10.1016/j.neuroscience.2009.12.020. Epub 2009 Dec 28. PMID 20036321
- [Background] Noda H, Takeuchi H, Mizuno T, Suzumura A. Fingolimod phosphate promotes the neuroprotective effects of microglia. J Neuroimmunol. 2013 Mar 15;256(1-2):13-8. doi: 10.1016/j.jneuroim.2012.12.005. Epub 2013 Jan 3. PMID 23290828
- [Background] Rothhammer V, Kenison JE, Tjon E, Takenaka MC, de Lima KA, Borucki DM, Chao CC, Wilz A, Blain M, Healy L, Antel J, Quintana FJ. Sphingosine 1-phosphate receptor modulation suppresses pathogenic astrocyte activation and chronic progressive CNS inflammation. Proc Natl Acad Sci U S A. 2017 Feb 21;114(8):2012-2017. doi: 10.1073/pnas.1615413114. Epub 2017 Feb 6. PMID 28167760
- [Background] Qin C, Fan WH, Liu Q, Shang K, Murugan M, Wu LJ, Wang W, Tian DS. Fingolimod Protects Against Ischemic White Matter Damage by Modulating Microglia Toward M2 Polarization via STAT3 Pathway. Stroke. 2017 Dec;48(12):3336-3346. doi: 10.1161/STROKEAHA.117.018505. Epub 2017 Nov 7. PMID 29114096
- [Background] Das A, Arifuzzaman S, Kim SH, Lee YS, Jung KH, Chai YG. FTY720 (fingolimod) regulates key target genes essential for inflammation in microglial cells as defined by high-resolution mRNA sequencing. Neuropharmacology. 2017 Jun;119:1-14. doi: 10.1016/j.neuropharm.2017.03.034. Epub 2017 Mar 31. PMID 28373076
- [Background] Sucksdorff M, Rissanen E, Tuisku J, Nuutinen S, Paavilainen T, Rokka J, Rinne J, Airas L. Evaluation of the Effect of Fingolimod Treatment on Microglial Activation Using Serial PET Imaging in Multiple Sclerosis. J Nucl Med. 2017 Oct;58(10):1646-1651. doi: 10.2967/jnumed.116.183020. Epub 2017 Mar 23. PMID 28336784
- [Background] Delbridge MS, Shrestha BM, Raftery AT, El Nahas AM, Haylor JL. Reduction of ischemia-reperfusion injury in the rat kidney by FTY720, a synthetic derivative of sphingosine. Transplantation. 2007 Jul 27;84(2):187-95. doi: 10.1097/01.tp.0000269794.74990.da. PMID 17667810
- [Background] Man K, Ng KT, Lee TK, Lo CM, Sun CK, Li XL, Zhao Y, Ho JW, Fan ST. FTY720 attenuates hepatic ischemia-reperfusion injury in normal and cirrhotic livers. Am J Transplant. 2005 Jan;5(1):40-9. doi: 10.1111/j.1600-6143.2004.00642.x. PMID 15636610
- [Background] Hasegawa Y, Suzuki H, Sozen T, Rolland W, Zhang JH. Activation of sphingosine 1-phosphate receptor-1 by FTY720 is neuroprotective after ischemic stroke in rats. Stroke. 2010 Feb;41(2):368-74. doi: 10.1161/STROKEAHA.109.568899. Epub 2009 Nov 25. PMID 19940275
- [Background] Wei Y, Yemisci M, Kim HH, Yung LM, Shin HK, Hwang SK, Guo S, Qin T, Alsharif N, Brinkmann V, Liao JK, Lo EH, Waeber C. Fingolimod provides long-term protection in rodent models of cerebral ischemia. Ann Neurol. 2011 Jan;69(1):119-29. doi: 10.1002/ana.22186. Epub 2010 Nov 12. PMID 21280082
- [Background] Fu Y, Zhang N, Ren L, Yan Y, Sun N, Li YJ, Han W, Xue R, Liu Q, Hao J, Yu C, Shi FD. Impact of an immune modulator fingolimod on acute ischemic stroke. Proc Natl Acad Sci U S A. 2014 Dec 23;111(51):18315-20. doi: 10.1073/pnas.1416166111. Epub 2014 Dec 8. PMID 25489101
- [Background] Zhu Z, Fu Y, Tian D, Sun N, Han W, Chang G, Dong Y, Xu X, Liu Q, Huang D, Shi FD. Combination of the Immune Modulator Fingolimod With Alteplase in Acute Ischemic Stroke: A Pilot Trial. Circulation. 2015 Sep 22;132(12):1104-1112. doi: 10.1161/CIRCULATIONAHA.115.016371. Epub 2015 Jul 22. PMID 26202811
- [Background] Lu L, Barfejani AH, Qin T, Dong Q, Ayata C, Waeber C. Fingolimod exerts neuroprotective effects in a mouse model of intracerebral hemorrhage. Brain Res. 2014 Mar 25;1555:89-96. doi: 10.1016/j.brainres.2014.01.048. Epub 2014 Feb 3. PMID 24502984
- [Background] Rolland WB, Lekic T, Krafft PR, Hasegawa Y, Altay O, Hartman R, Ostrowski R, Manaenko A, Tang J, Zhang JH. Fingolimod reduces cerebral lymphocyte infiltration in experimental models of rodent intracerebral hemorrhage. Exp Neurol. 2013 Mar;241:45-55. doi: 10.1016/j.expneurol.2012.12.009. Epub 2012 Dec 21. PMID 23261767
- [Background] Sun N, Shen Y, Han W, Shi K, Wood K, Fu Y, Hao J, Liu Q, Sheth KN, Huang D, Shi FD. Selective Sphingosine-1-Phosphate Receptor 1 Modulation Attenuates Experimental Intracerebral Hemorrhage. Stroke. 2016 Jul;47(7):1899-906. doi: 10.1161/STROKEAHA.115.012236. Epub 2016 May 12. PMID 27174529
- [Background] Fu Y, Hao J, Zhang N, Ren L, Sun N, Li YJ, Yan Y, Huang D, Yu C, Shi FD. Fingolimod for the treatment of intracerebral hemorrhage: a 2-arm proof-of-concept study. JAMA Neurol. 2014 Sep;71(9):1092-101. doi: 10.1001/jamaneurol.2014.1065. PMID 25003359
- [Background] Murthy SB, Moradiya Y, Shah J, Merkler AE, Mangat HS, Iadacola C, Hanley DF, Kamel H, Ziai WC. Nosocomial Infections and Outcomes after Intracerebral Hemorrhage: A Population-Based Study. Neurocrit Care. 2016 Oct;25(2):178-84. doi: 10.1007/s12028-016-0282-6. PMID 27350549
- [Background] Lord AS, Gilmore E, Choi HA, Mayer SA; VISTA-ICH Collaboration. Time course and predictors of neurological deterioration after intracerebral hemorrhage. Stroke. 2015 Mar;46(3):647-52. doi: 10.1161/STROKEAHA.114.007704. Epub 2015 Feb 5. PMID 25657190
- [Background] Dobin A, Davis CA, Schlesinger F, Drenkow J, Zaleski C, Jha S, Batut P, Chaisson M, Gingeras TR. STAR: ultrafast universal RNA-seq aligner. Bioinformatics. 2013 Jan 1;29(1):15-21. doi: 10.1093/bioinformatics/bts635. Epub 2012 Oct 25. PMID 23104886
- [Background] Liao Y, Smyth GK, Shi W. featureCounts: an efficient general purpose program for assigning sequence reads to genomic features. Bioinformatics. 2014 Apr 1;30(7):923-30. doi: 10.1093/bioinformatics/btt656. Epub 2013 Nov 13. PMID 24227677
- [Background] Love MI, Huber W, Anders S. Moderated estimation of fold change and dispersion for RNA-seq data with DESeq2. Genome Biol. 2014;15(12):550. doi: 10.1186/s13059-014-0550-8. PMID 25516281
- [Background] Ching T, Huang S, Garmire LX. Power analysis and sample size estimation for RNA-Seq differential expression. RNA. 2014 Nov;20(11):1684-96. doi: 10.1261/rna.046011.114. Epub 2014 Sep 22. PMID 25246651
- [Background] Benjamini Y, Hochberg Y. Controlling the False Discovery Rate: A Practical and Powerful Approach to Multiple Testing. Journal of the Royal Statistical Society Series B (Methodological). 1995;57(1):289-300
- [Background] Kramer A, Green J, Pollard J Jr, Tugendreich S. Causal analysis approaches in Ingenuity Pathway Analysis. Bioinformatics. 2014 Feb 15;30(4):523-30. doi: 10.1093/bioinformatics/btt703. Epub 2013 Dec 13. PMID 24336805
- [Background] Huang DW, Sherman BT, Tan Q, Kir J, Liu D, Bryant D, Guo Y, Stephens R, Baseler MW, Lane HC, Lempicki RA. DAVID Bioinformatics Resources: expanded annotation database and novel algorithms to better extract biology from large gene lists. Nucleic Acids Res. 2007 Jul;35(Web Server issue):W169-75. doi: 10.1093/nar/gkm415. Epub 2007 Jun 18. PMID 17576678
- See also: Minimally Invasive Surgery Plus Rt-PA for ICH Evacuation Phase III — https://ClinicalTrials.gov/show/NCT01827046
- See also: MIND: Artemis in the Removal of Intracerebral Hemorrhage — https://ClinicalTrials.gov/show/NCT03342664
- See also: ENRICH: Early MiNimally-invasive Removal of IntraCerebral Hemorrhage (ICH) — https://ClinicalTrials.gov/show/NCT02880878

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients coming the Emergency Department or direct admitted to the Neurosciences Intensive Care Unit at Wake Forest Baptist Hospital between August 2020 and June 2023 with the diagnosis of spontaneous ICH will be identified as potentially eligible participants and screened by interview.
Pre-assignment Details: Consented participants who can be administered an oral drug will be allocated to Fingolimod or Placebo study groups using a computer-based random number-generating allocation. Consented participants who are unable to be administered the oral drug or placebo are assigned to the open-label group.
Groups:
- Control: In addition to Standard of care treatment, those participants randomized to the control group will receive a single dose placebo pill within 24 hours of symptom onset
  Control: A single oral placebo pill within 24 hours of symptom onset
- Open-label Fingolimod: In addition to standard of care treatment,10 subjects will be assigned to the open-label group who will receive a single dose of 0.5 mg oral fingolimod within 24 hours of symptom onset to assess feasibility of administration through NGT or Dobhoff tube.
  Open-label Fingolimod: A single dose of 0.5 mg fingolimod through an NGT or Dobhoff tube within 24 hours of symptom onset
Period: Overall Study
Arm/Group | Fingolimod | Control | Open-label Fingolimod
Started (Enrollment) | 9 | 8 | 11
24h Post-ictus | 8 | 7 | 11
72h Post-ictus | 9 | 7 | 10
5-7 Days | 9 | 6 | 7
10-14 Days | 4 | 2 | 7
30 Days | 9 | 5 | 7
90 Days | 9 | 5 | 8
180 Days | 6 | 5 | 5
365 Days | 3 | 4 | 6
Completed | 3 | 4 | 3
Not Completed | 6 | 4 | 8
Not completed — Lost to Follow-up | 3 | 2 | 6
Not completed — Death | 3 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fingolimod | Control | Open-label Fingolimod | Total
Number analyzed (Participants) | 9 | 8 | 11 | 28
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71.0 [67.0 to 77.0] | 67.0 [64.8 to 69.0] | 59.0 [48.5 to 67.5] | 66.0 [54.8 to 74.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 6 | 10
  Male | 7 | 6 | 5 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 4 | 7
  Not Hispanic or Latino | 8 | 6 | 7 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 6
  White | 7 | 6 | 9 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Prior stroke [Count of Participants; unit: Participants] | 0 | 2 | 1 | 3
Hypertension [Count of Participants; unit: Participants] | 5 | 8 | 8 | 21
Diabetes [Count of Participants; unit: Participants] | 2 | 0 | 4 | 6
Coronary Artery Disease [Count of Participants; unit: Participants] | 1 | 2 | 2 | 5
Hyperlipidemia [Count of Participants; unit: Participants] | 3 | 4 | 4 | 11
Obesity [Count of Participants; unit: Participants] | 0 | 2 | 3 | 5
Atrial Fibrillation [Count of Participants; unit: Participants] | 2 | 1 | 1 | 4
Smoking Status [Count of Participants; unit: Participants]
  Current or Former | 4 | 4 | 3 | 11
  Never | 4 | 1 | 5 | 10
  Unknown | 1 | 3 | 3 | 7
Antiplatelet medication [Count of Participants; unit: Participants] | 3 | 3 | 2 | 8
Anticoagulant Medication [Count of Participants; unit: Participants] | 4 | 2 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Cardiac Events
Description: Number of participants with clinically significant cardiac events. Clinically significant cardiac events include myocardial infarction, unstable angina, stroke, transient ischemic attack, any heart failure, bradycardia and heart block. Cardiac events were monitored with telemetry up to and after 72 hours while hospitalized. A check in was performed at 30 days with an in-person clinical or hospital visit to ascertain any cardiac events via patient discussion and medical record review.
Time Frame: up to 30 days post-ictus
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Fingolimod | Control | Open-label Fingolimod
Number analyzed (Participants) | 9 | 8 | 11
Participants | 3 | 0 | 0
Statistical Analysis 1: Comparison: Fingolimod vs Control vs Open-label Fingolimod; Difference in proportion of subjects with cardiac events up to 30 days post-ictus tested between three groups; Test type: Superiority; p = 0.0427, Fisher Exact — p<0.05 considered significant. Between group pairwise comparisons performed with Bonferroni correction

2. Primary Outcome: Rate of Nosocomial Infections (UTI, Sepsis, and Pneumonia)
Description: Rate of nosocomial infections (UTI, sepsis, and pneumonia) by group
Time Frame: up to 90 days post-ictus
Population: All enrolled participants by group
Measure: Count of Participants; unit: Participants
Arm/Group | Fingolimod | Control | Open-label Fingolimod
Number analyzed (Participants) | 9 | 8 | 11
Participants | 1 | 1 | 5
Statistical Analysis 1: Comparison: Fingolimod vs Control vs Open-label Fingolimod; Difference in proportion of subjects with nosocomial infections up to 90 days post-ictus tested between three groups. No pairwise comparisons performed; Test type: Superiority; p = 0.19, Fisher Exact

3. Primary Outcome: Rate of Neurologic Decline
Description: considered a change ≥ 4 points of the NIHSS between enrollment and 30 days post-ictus. A higher score indicates higher severity and poorer prognosis. Scale is 0-42.
Time Frame: up to 30 days post-ictus
Population: All three arms where data were available at 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fingolimod | Control | Open-label Fingolimod
Number analyzed (Participants) | 7 | 5 | 7
Participants | 2 | 0 | 0
Statistical Analysis 1: Comparison: Fingolimod vs Control vs Open-label Fingolimod; Difference in proportion of subjects with neurologic decline up to 30 days post-ictus tested between three groups. No pairwise comparisons performed; Test type: Superiority; p = 0.30, Fisher Exact

4. Secondary Outcome: Rate of Successful Administration of Fingolimod Through an NGT or Dobhoff Tube
Description: Rate of successful administration of fingolimod through an NGT or Dobhoff tube in Open-label group only
Time Frame: Enrollment
Population: 11 subjects enrolled in open-label arm
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Fingolimod
Number analyzed (Participants) | 11
Participants | 11

5. Secondary Outcome: Percent Change in Lymphocyte Subpopulations of CD4+ T Cells
Description: Percent Change in Lymphocyte Subpopulations of CD4+ T Cells
Time Frame: Enrollment to 30 days
Population: Subjects where 30 day labs were obtained are included in this analysis
Measure: Median (Full Range); unit: percent change
Arm/Group | Fingolimod | Control | Open-label Fingolimod
Number analyzed (Participants) | 6 | 4 | 6
percent change | 19.6 [-18.8 to 81.9] | -2.56 [-10.3 to 3.52] | -5.00 [-14.7 to 40.5]

6. Secondary Outcome: Percent Change in Lymphocyte Subpopulations of CD8+ T Cells
Description: Percent change in lymphocyte subpopulations of CD8+ T Cells
Time Frame: Enrollment and 30 days
Population: Subjects where 30 day labs were obtained are included in this analysis
Measure: Median (Full Range); unit: percent change
Arm/Group | Fingolimod | Control | Open-label Fingolimod
Number analyzed (Participants) | 6 | 4 | 6
percent change | 19.3 [-20.4 to 59.0] | 21.4 [-6.09 to 113] | 21.6 [-61.5 to 82.9]

7. Secondary Outcome: Percent Change in Lymphocyte Subpopulations of CD19+ B Cells
Description: Percent change in lymphocyte subpopulations of CD19+ B cells
Time Frame: Enrollment and 30 days
Population: Subjects where 30 day labs were obtained are included in this analysis
Measure: Median (Full Range); unit: percent change
Arm/Group | Fingolimod | Control | Open-label Fingolimod
Number analyzed (Participants) | 6 | 4 | 6
percent change | 121 [-39.4 to 186] | 0.230 [-16.9 to 16.5] | 9.22 [-84.1 to 43.8]

8. Secondary Outcome: Change in Hematoma Volume Obtained by MRI
Description: Average decrease per day by group in volumetric measurement calculations of hematoma obtained by MRI between enrollment and 365 days. All MRI imaging data obtained on hematoma volume between enrollment and 365 days were used to calculate estimates via a linear mixed effects model controlling for repeated measures within subject.
Time Frame: Enrollment and 365 days
Population: All enrolled subjects included in analysis. Fingolimod group included 18 observations, placebo included 14 observations and open-label included 23 observations across the time period.
Measure: Mean (Standard Error); unit: mm^3 per day
Arm/Group | Fingolimod | Control | Open-label Fingolimod
Number analyzed (Participants) | 9 | 8 | 11
mm^3 per day | -247.19 (75.68) | -86.29 (17.74) | -210.03 (23.81)

9. Secondary Outcome: Change in Hematoma Volume Obtained by CT
Description: Average decrease per day by group in volumetric measurement calculations of hematoma obtained by CT between enrollment and 365 days. All CT imaging data obtained on hematoma volume between enrollment and 365 days were used to calculate estimates via a linear mixed effects model controlling for repeated measures within subject.
Time Frame: Enrollment and 365 days
Population: All enrolled subjects included in analysis. Fingolimod group included 46 observations, placebo included 39 observations and open-label included 60 observations across the time period.
Measure: Mean (Standard Error); unit: mm^3 per day
Arm/Group | Fingolimod | Control | Open-label Fingolimod
Number analyzed (Participants) | 9 | 8 | 11
mm^3 per day | -156.84 (46.35) | -90.56 (54.89) | -86.73 (15.95)

10. Secondary Outcome: Change in Peri-hematomal Edema Volume Obtained by CT
Description: Average decrease per day by group in volumetric measurement calculations of peri-hematomal edema volume between enrollment and 365 days. All CT imaging data obtained on peri-hematomal edema volume between enrollment and 365 days were used to calculate estimates via a linear mixed effects model controlling for repeated measures within subject.
Time Frame: Enrollment to 365 days
Population: as for outcome 9
Measure: Mean (Standard Error); unit: mm^3
Arm/Group | Fingolimod | Control | Open-label Fingolimod
Number analyzed (Participants) | 9 | 8 | 11
mm^3 | -65.85 (47.50) | -62.21 (64.76) | -64.93 (16.33)

11. Secondary Outcome: Change in Peri-hematomal Edema Volume Obtained by MRI
Description: Average decrease per day by group in volumetric measurement calculations of peri-hematomal edema obtained from radiographic imaging (MRI) between enrollment and 365 days. All MRI imaging data obtained on peri-hematomal edema volume between enrollment and 365 days were used to calculate estimates via a linear mixed effects model controlling for repeated measures within subject.
Time Frame: Enrollment to 365 days
Population: as for outcome 8
Measure: Mean (Standard Error); unit: mm^3
Arm/Group | Fingolimod | Control | Open-label Fingolimod
Number analyzed (Participants) | 9 | 8 | 11
mm^3 | -327.12 (89.61) | -118.36 (31.75) | -74.96 (55.84)

12. Secondary Outcome: National Institutes of Health Stroke Scale Total Score (NIHSS)
Description: The scoring range is 0 to 42 points, with higher numbers indicating greater severity. (NIHSS)
Time Frame: 365 days
Population: Subjects where score was collected at 365 days.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Fingolimod | Control | Open-label Fingolimod
Number analyzed (Participants) | 2 | 4 | 4
score on a scale | 0 [0 to 0] | 1 [1 to 2] | 5 [0 to 8]

13. Secondary Outcome: Interviewer-administered Modified Rankin Scale (mRS)
Description: The modified Rankin Scale (mRS) will measure functional recovery and ability to perform activities of daily living. The mRS is a 6 point disability scale with scores ranging from 0 (no symptoms) to 5 (severe disability) with 6 indicating death. Lower scores denote better outcome.
Time Frame: 365 days post-ictus
Population: Subjects where scores were collected at 365 days.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Fingolimod | Control | Open-label Fingolimod
Number analyzed (Participants) | 2 | 4 | 6
score on a scale | 1.5 [1 to 2] | 1.5 [1 to 2] | 2.5 [1 to 3]

14. Secondary Outcome: Patient-Reported Outcomes Measurement Information (PROMIS) 10 Questionnaire
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) 10 questionnaire will measure patient self-reporting of physical and neurobehavioral functions. Mean T-score for general population is 50 with standard deviation of 10. Higher T-scores indicate better physical and mental health. Typically, T-score ranges from 20 to 80.
Time Frame: 365 days
Population: Subjects completing instrument at 365 days.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Fingolimod | Control | Open-label Fingolimod
Number analyzed (Participants) | 2 | 4 | 3
score on a scale
  Physical T Score | 48.2 [42.3 to 54.1] | 55.9 [44.9 to 61.9] | 47.7 [39.8 to 50.8]
  Mental T Score | 53.4 [47.7 to 59.0] | 47.7 [33.8 to 62.5] | 41.1 [41.1 to 50.8]

15. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: Montreal Cognitive Assessment (MoCA) will measure recovery (neurocognitive). Scores range from 0 to 30 with higher scores denoting better outcomes.
Time Frame: 365 days
Population: Subjects completing instrument at 365 days.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Fingolimod | Control | Open-label Fingolimod
Number analyzed (Participants) | 2 | 4 | 3
score on a scale | 25 [24 to 26] | 24 [21 to 25] | 20 [17 to 25]

16. Secondary Outcome: Western Aphasia Battery-Revised (WAB-R)
Description: Western Aphasia Battery-Revised (WAB-R) will measure recovery (neurocognitive and speech). Language and Aphasia subscale scores both range from 0 to 100. Higher scores denote better outcome.
Time Frame: 365 days
Population: Subjects completing instrument at 365 days.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Fingolimod | Control | Open-label Fingolimod
Number analyzed (Participants) | 2 | 4 | 3
score on a scale
  Language score | 98.8 [97.5 to 100] | 96.9 [86.9 to 98.8] | 90.0 [70.6 to 93.1]
  Aphasia score | 100 [100 to 100] | 98.3 [94.2 to 100] | 95.0 [73.3 to 95.8]

17. Secondary Outcome: Mortality
Description: Mortality at 30 days
Time Frame: 30 days
Population: All enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Fingolimod | Control | Open-label Fingolimod
Number analyzed (Participants) | 9 | 8 | 11
Participants | 0 | 1 | 0

18. Secondary Outcome: Mortality
Description: Mortality at 90 days
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fingolimod | Control | Open-label Fingolimod
Number analyzed (Participants) | 9 | 8 | 11
Participants | 1 | 1 | 0

19. Secondary Outcome: All Cause Mortality
Description: All cause mortality within 365 days
Time Frame: up to 365 days
Population: All enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Fingolimod | Control | Open-label Fingolimod
Number analyzed (Participants) | 9 | 8 | 11
Participants | 3 | 1 | 1

ADVERSE EVENTS:
Time Frame: Enrollment to 365 days
Arm/Group | Fingolimod | Control | Open-label Fingolimod
All-Cause Mortality (participants affected / at risk) | 3/9 | 1/8 | 1/11
Serious Adverse Events (participants affected / at risk) | 3/9 | 1/8 | 5/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fingolimod (N=9) | Control (N=8) | Open-label Fingolimod (N=11)
Cardiac event (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT04088630/Prot_SAP_001.pdf
  • Informed Consent Form (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT04088630/ICF_000.pdf